CLINICAL TRIAL: NCT05759455
Title: Vitamen D in Autism
Brief Title: Assessment of Vitamin D Level in Children With Autism in Assiut University Children Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelmoneim Ahmed, assiutU, Assiut University
Other Study IDs: vitamin d in autism
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Assessment of Vitamin D Level in Children With Autism in Assiut University Children Hospital
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: vitamin d — Assessment of Vitamin D level in Children with Autism in assiut university children hospital

SUMMARY:
In the present study, we aim to evaluate the serum level of 25 hydrxy vitamin D in autistic children .

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a group of neurodevelopmental disorders characterized by impaired social interaction and communication, repetitive and stereotyped behaviors, and restricted interests ( Lord et al,2018).

Autism is becoming increasingly common. Recently, the Centers for Disease Control and Prevention reported that the prevalence of autism among 8-year-old children in the United States in 2016 was 1/54, with a 4.3:1 ratio of males to females ( Maenner et al ,2020).

Autistic individuals manifest problematic behaviors, such as attacking, self-injury, resistance to orders, and failure of normal conversation, and are usually comorbid with social-anxiety, attention-deficit/hyperactivity, sleep-wake disorders, and obsessive-compulsive disorders. As such, it is difficult for them to obtain the same education levels as their neurotypical peers, find full-time jobs, or live independently ( Lord et al,2018),( Lai et al , 2019) .

Fortunately, evidence indicates that appropriate and early intervention could help autistic individuals improve their symptoms and life quality (Landa ., 2018).

Notably, research shows that nutritional and dietary intervention is an effective way to improve nutritional status, non-verbal IQ, and autism symptoms (Adams et al ,2018). Therefore, it is essential to identify physiological dysfunction and abnormal nutritional status in autistic individuals and then take corresponding interventions.

Autism is a multifactorial disorder resulting from an interaction of genetic and environmental factors. Hundreds of autism risk genes and various environmental factors have been discovered ( Linhong et al 2020) ( Lord et al , 2020). Possible environmental factors include folic acid deficiency, neonatal hypoxia, maternal obesity, and gestational diabetes mellitus( Lord et al , 2020).

Recently, emerging evidence suggests that vitamin D deficiency might be an unfavorable factor of autism (Mazahery et al, 2016).

Vitamin D is a steroid hormone; it is primarily synthesized in the skin under UV-B light, and a small amount is derived from dietary intake (Saraff et al , 2016).

Although the underlying mechanisms between vitamin D and autism are unclear, there is some biological evidence indicating the potential link. Vitamin D-metabolizing enzymes and vitamin D receptors are widely expressed in immune cells, the placenta, and the developing and adult brain; high levels of vitamin D surface receptor (protein disulfide isomerase family A members 3, PDIA3) are found in the cortex and hippocampus, which suggests the association between vitamin D, and brain development and function (Bivona G., et al, 2019)( Landel et al, 2018)( Wang et al, 2012).

Indeed, vitamin D has important effects on brain development and function, including neuronal differentiation, proliferation and apoptosis, regulating synaptic plasticity, the ontogeny of the dopaminergic system, immunomodulation, and reducing oxidative burden (Bivona et al, 2019).

In addition, vitamin D plays an important role in the regulation of gene expression. One study showed that 223 ASD risk genes in the SFARI database were vitamin D3-sensitive genes, which meant that these ASD related genes might be regulated by vitamin D (Trifonova et al, 2019).

ELIGIBILITY:
Inclusion Criteria:

* Patient who full filled the diagnostic criteria of autism spectrum disorder according to DSM-IV.

Exclusion Criteria:

* 1)Children using vitamin D supplement. 2)patients with associated congenital malformation. 3)patients with chromosomal abnormalities. 4)patients with chronic physical illness. 5)patients with epilepsy. 6)patients with hepatic or renal disease.

Ages: 10 Months to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: 1. full history.
  2. full clinical examination.
  3. diagnosis of patients with ASD based on medical experience,clinical examination and two criteria of DSM-IV .
  4. evaluation of serum 25 hydroxy vitamin D level ; 5 ml of venous blood sample is taken for the test.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of Vitamin D level in Children with Autism in assiut university children hospital | 2 years
  In the present study, we aim to evaluate the serum level of 25 hydrxy vitamin D in autistic children .

REFERENCES:
- See also: 1.Adams J., Audhya T., Matthews J.S., Li K., Naviaux J.C., Naviaux R.K., Adams R.L., Coleman D.M., Quig D.W., Geis E., et al. Comprehensive Nutritional and Dietary Intervention for Autism Spectrum Disorder — https://pubmed.ncbi.nlm.nih.gov/17356557/